CLINICAL TRIAL: NCT02642796
Title: Comparison of the Efficacy of Two Different Transcutaneous Electrical Nerve Stimulation Application Sites in Reducing Postoperative Pain After Hip Fracture Surgery
Brief Title: Transcutaneous Nerve Stimulation for Post-operative Acute and Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, MENEKSE OKSAR, Assistant Professor, Mustafa Kemal University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2013/34
Record Dates: First submitted 2015-12-25; First posted 2015-12-30 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain; Hip Fracture
Keywords: Percutaneous Electric Nerve Stimulation; Lumbosacral plexus; surgical wound; postoperative analgesia; transcutaneous electrical stimulation
MeSH Terms: conditions — Pain, Postoperative; Hip Fractures; Surgical Wound | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I (control) (No Intervention): Patient controlled analgesia (epidural fentanyl): PCA only
- group II (Experimental): PCA plus lumbar plexus & sciatic nerve transcutaneous electric nerve stimulation (LS-TENS)
  Interventions: Device: transcutaneous electric nerve stimulation
- group III (Experimental): PCA plus surgical wound transcutaneous electric nerve stimulation ( SW-TENS)
  Interventions: Device: transcutaneous electric nerve stimulation

INTERVENTIONS:
Device: transcutaneous electric nerve stimulation — The TENS device will be applied for treatment periods of 30-40 minutes. The electrodes will be connected to the TENS device are stimulated in modulation mode and the parameters will be adjusted as pulse width of 60 μs,frequency of 120 Hz and the stimulation intensity as high as the subject could tolerate.
  Electrodes will be placed on either lumbar and sciatic nerve tracing unilaterally or on either side or parallel to the surgical wound.
  Other Names: Intelect portable TENS
  Arms: group II; group III

SUMMARY:
Aim of the study to assess the efficacy of two modes of transcutaneous electrical nerve stimulation (TENS) on relief of postoperative acute pain after hip fracture surgery.

DETAILED DESCRIPTION:
The patients underwent undergo fractured hip surgery will be distributed into three groups with respect to the mode of postoperative analgesia applied: Group I (control): PCA only; group II: PCA plus lumbar plexus & sciatic nerve TENS (LS-TENS); group III: PCA plus surgical wound TENS (SW-TENS). TENS will be applied every 2 hours for 30-40 minutes during 48 hours postoperatively. Visual analogue score (VAS), Ramsey sedation scores, frequencies of PCA demand and counts of PCA delivery, as well as total analgesic consumption will be noted and compared between groups at various time intervals.

Visual analog scale (VAS) will be applied at 2 months postoperatively VAS and Mcgill pain questionnaire will be applied at the 6th and 24th months of the surgery to assess acute and chronic pain in the study population and the differences among groups.

ELIGIBILITY:
Inclusion Criteria: Adult patients will be scheduled for surgery due to hip fracture in Mustafa Kemal University Hospital will be included in the study.

Exclusion Criteria: Patients with a history of opioid analgesic abuse, or sensitivity to opioids, and those with clinically significant systemic (cardiovascular, pulmonary, hepatic, renal, neurologic etc.) diseases, will be excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Visual analog scale for pain | 48 h postoperatively
  Postoperative pain intensity is assessed using VAS for pain postoperatively.

SECONDARY OUTCOMES:
Ramsey sedation scores | 48 h postoperatively
  Sedation score is assessed for safety of epidural analgesic use.
Frequencies of PCA demand | 48 h postoperatively
  Patient demand will be assessed by PCA demand
PCA delivery counts | 48 h postoperatively
  Delivery count shows the actual PCA delivery. It is different from the demand.
Total fentanyl consumption | 48 h postoperatively
  Total analgesic use during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Menekse Oksar, M.D., Principal Investigator — Mustafa Kemal University Medical School
Locations (1):
- Mustafa Kemal University Hospital, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hamza MA, White PF, Ahmed HE, Ghoname EA. Effect of the frequency of transcutaneous electrical nerve stimulation on the postoperative opioid analgesic requirement and recovery profile. Anesthesiology. 1999 Nov;91(5):1232-8. doi: 10.1097/00000542-199911000-00012. PMID 10551571
- [Result] Wang B, Tang J, White PF, Naruse R, Sloninsky A, Kariger R, Gold J, Wender RH. Effect of the intensity of transcutaneous acupoint electrical stimulation on the postoperative analgesic requirement. Anesth Analg. 1997 Aug;85(2):406-13. doi: 10.1097/00000539-199708000-00029. PMID 9249122
- [Result] Lan F, Ma YH, Xue JX, Wang TL, Ma DQ. Transcutaneous electrical nerve stimulation on acupoints reduces fentanyl requirement for postoperative pain relief after total hip arthroplasty in elderly patients. Minerva Anestesiol. 2012 Aug;78(8):887-95. Epub 2012 Apr 24. PMID 22531569
- [Derived] Oksar M, Kalaci A, Turhanoglu S. Transcutaneous electrical nerve stimulation for reducing postoperative acute pain after hip fracture surgery: a double-blinded randomized clinical trial. Eur Rev Med Pharmacol Sci. 2024 Apr;28(7):2788-2796. doi: 10.26355/eurrev_202404_35907. PMID 38639518
- See also: Use of TENS at mixed (2- and 100-Hz) frequencies of stimulation produced a slightly greater opioid-sparing effect than either low (2-Hz) or high (100 Hz) frequencies alone. — http://www.ncbi.nlm.nih.gov/pubmed/10551571
- See also: High-TAES (9-12 mA) produced a significant decrease in the PCA opioid requirement and opioid-related side effects after low intraabdominal surgery. — http://www.ncbi.nlm.nih.gov/pubmed/9249122
- See also: TENS on specific acupoints is an effective and complementary approach to reduce postoperative analgesic requirement in elderly patients after total hip arthroplasty.. — http://www.ncbi.nlm.nih.gov/pubmed/?term=Transcutaneous+electrical+nevre+stimulation+on+acupoints+reduces+fentanyl+requirement+for+postoperative+pain+relief+after+total+hiparthroplasty+in